CLINICAL TRIAL: NCT03952702
Title: The Long-Term Efficacy of Overminus Lens Therapy in Intermittent Exotropia
Brief Title: Overminus Lens Therapy in Intermittent
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Elif Demirkilinc Biler, Assoc. Prof., M.D., Ege University
Other Study IDs: Ege30042919
Record Dates: First submitted 2019-04-30; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Intermittent Exotropia; Myopia Overcorrection; Over-minus Therapy; Myopia Progression
Keywords: Intermittent exotropia; overminus lens therapy; myopic overcorrection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Myopic overcorrection — Myopic overcorrection

SUMMARY:
In this prospective study, entitled "The Long-Term Efficacy of Overminus Lens Therapy in Intermittent Exotropia",the investigators examined the long-term impact of overminus lenses on the management of intermittent exotropia (IXT), treatment effect after overminus treatment has been discontinued and also investigated if overminus lenses cause myopia in long-term.

DETAILED DESCRIPTION:
Purpose: To evaluate the long-term impact of overminus lenses in intermittent exotropia (IXT), to determine if the treatment effect would persist after overminus minus lenses are discontinued and also to investigate if overminus lenses cause myopia.

Materials and Method: Sixty-five consecutive cases of IXT followed for at least 48 months were included. Patients with a history of previous surgery, ocular pathology, convergence insufficiency, severe myopia (>-5.0 D), severe hyperopia (>+5.0 D), moderate or severe amblyopia and poor compliance with spectacles were excluded. Data was collected including near stereoacuity, AC/A ratio, control of IXT measured with Newcastle Control Score (NCS) at baseline and in all follow-up visits. Baseline values without overminus threapy were compared with postintervention values at every visit.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with IXT
* prescribed overminus lenses

Exclusion Criteria:

* a history of previous surgery, ocular pathology
* convergence insufficiency type IXT
* presence of any type of ocular deviation except IXT
* presence of severe myopia (greater than -5.0 D)
* presence of severe hyperopia (greater than +5.0 D)
* presence of moderate or severe amblyopia
* poor compliance with overminus spectacles
* follow up period of <48 months after intervention.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All consecutive pediatric patients diagnosed with IXT and prescribed overminus lenses
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
The long-term effect of overminus lenses in fusional capacity of patients with intermittent exotropia. | 4 years
  Overminus lenses were prescribed on the treatment of intermittent exotropia as the first choice. To investigate the effect of overminus lenses on treatment, progress in fusional capability of the patients evaluated with Newcastle control score system were investigated.
The long-term effect of overminus lenses on stereopsis of patients with intermittent exotropia. | 4 years
  Changes in stereopsis values (arcsec) evaluated with TNO test were observed.
The long-term effect of prescribing overminus lenses on refractive changes. | 4 years
  Refractive data of the patients in terms of dioptri were measured with autorefractometer during the long-term follow-up period to observe presence of any myopic shift.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No